CLINICAL TRIAL: NCT01553747
Title: A Randomized, Double-blind, Placebo-controlled, Phase 3 Study to Evaluate the Efficacy, Safety, and Tolerability of JNJ-27018966 in the Treatment of Patients With Diarrhea-Predominant Irritable Bowel Syndrome
Brief Title: Efficacy, Safety, and Tolerability of Eluxadoline in the Treatment of Participants With Diarrhea-Predominant Irritable Bowel Syndrome (IBS-d)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Furiex Pharmaceuticals, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 27018966IBS3002; 2012-001601-24 (EudraCT Number)
Record Dates: First submitted 2012-03-08; First posted 2012-03-14 (Estimated); Results first posted 2018-07-30 (Actual); Last update posted 2018-07-30 (Actual); Status verified 2018-07

CONDITIONS: Irritable Bowel Syndrome
Keywords: Irritable bowel syndrome with diarrhea; Irritable bowel syndrome; Diarrhea predominant irritable bowel syndrome; Colonic diseases; Colonic diseases, functional; Digestive system disease; Gastrointestinal disease; Intestinal disease; Colonic pseudo-obstruction; Diarrhea; Signs and symptoms, Digestive
MeSH Terms: conditions — Irritable Bowel Syndrome; Colonic Diseases; Colonic Diseases, Functional; Digestive System Diseases; Gastrointestinal Diseases; Intestinal Diseases; Colonic Pseudo-Obstruction; Diarrhea; Signs and Symptoms, Digestive | interventions — eluxadoline

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Eluxadoline 75 mg (Experimental): Eluxadoline 75 mg tablets, orally, twice daily for up to 26 weeks period.
  Interventions: Drug: Eluxadoline
- Eluxadoline 100 mg (Experimental): Eluxadoline 100 mg tablets, orally, twice daily for up to 26 weeks period.
  Interventions: Drug: Eluxadoline
- Placebo (Placebo Comparator): Eluxadoline placebo matching tablets, orally, twice daily for up to 26 weeks period.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Eluxadoline — Oral tablets twice daily
  Other Names: JNJ-27018966
  Arms: Eluxadoline 100 mg; Eluxadoline 75 mg
Drug: Placebo — Oral tablets twice daily
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine the efficacy, safety, and tolerability of different doses of eluxadoline (JNJ-27018966) compared with placebo in the treatment of participants with diarrhea-predominant irritable bowel syndrome.

ELIGIBILITY:
Inclusion Criteria:

1. Participant is 18 to 80 years old
2. Participant has a diagnosis of irritable bowel syndrome (IBS) with a subtype of diarrhea defined by the Rome III criteria.

2. Participant has had a colonoscopy performed:

* Within 10 years prior to Prescreening if participant is at least 50 years of age (sigmoidoscopy, double contrast barium enema, or computed tomography (CT) colonography within the past 5 years is acceptable)
* Since the onset (if applicable) of any of the following alarm features for participants of any age

  * Participant has documented weight loss within the past 6 months
  * Participant has nocturnal symptoms
  * Participant has a familial history of first-degree relatives with colon cancer
  * Participant has blood mixed with their stool (excluding blood from hemorrhoids).

    3. Female participants must be:
* Postmenopausal, defined as 52 years or older and amenorrheic for at least 2 years at Prescreening,
* Surgically sterile (have had a hysterectomy or bilateral oophorectomy, tubal ligation, or otherwise be incapable of pregnancy),
* Abstinent, or
* If sexually active, be practicing an effective method of birth control.

Exclusion Criteria:

1. Participant has a diagnosis of IBS with a subtype of constipation, mixed IBS, or unsubtyped IBS by the Rome III criteria.
2. Participant has a history of inflammatory or immune-mediated gastrointestinal (GI) disorders including inflammatory bowel disease (ie, Crohn's disease, ulcerative colitis) and celiac disease.
3. Participant has a history of diverticulitis within 3 months prior to Prescreening.
4. Participant has a history of intestinal obstruction, stricture, toxic megacolon, GI perforation, fecal impaction, gastric banding, bariatric surgery, adhesions, ischemic colitis, or impaired intestinal circulation (eg, aortoiliac disease).
5. Participant has any of the following surgical history:

   * Cholecystectomy with any history of post cholecystectomy biliary tract pain
   * Any abdominal surgery within the 3 months prior to Prescreening
   * Participant has a history of major gastric, hepatic, pancreatic, or intestinal surgery (appendectomy, hemorrhoidectomy, or polypectomy greater than 3 months post surgery are allowed)

Other protocol-specific eligibility criteria may apply.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1146 (Actual)
Dates: Start 2012-05-29 (Actual); Primary Completion 2014-01-09 (Actual); Study Completion 2014-01-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (213):
- United States (192):
  - Furiex Research Site, Birmingham, Alabama
  - Furiex Research Site, Decatur, Alabama
  - Furiex Research Site, Huntsville, Alabama
  - Furiex Research Site, Mobile, Alabama
  - Furiex Research Site, Montgomery, Alabama
  - Furiex Research Site, Sheffield, Alabama
  - Furiex Research Site, Tuscaloosa, Alabama
  - Furiex Research Site, Glendale, Arizona
  - Furiex Research Site, Mesa, Arizona
  - Furiex Research Site, Phoenix, Arizona
  - Furiex Research Site, Tucson, Arizona
  - Furiex Research Site, Jonesboro, Arkansas
  - Furiex Research Site, Little Rock, Arkansas
  - Furiex Research Site, Sherwood, Arkansas
  - Furiex Research Site, Anaheim, California
  - Furiex Research Site, Chula Vista, California
  - Furiex Research Site, Encinitas, California
  - Furiex Research Site, Garden Grove, California
  - Furiex Research Site, Huntington Beach, California
  - Furiex Research Site, Irvine, California
  - Furiex Research Site, La Mesa, California
  - Furiex Research Site, La Mirada, California
  - Furiex Research Site, Laguna Hills, California
  - Furiex Research Site, Lakewood, California
  - Furiex Research Site, Lincoln, California
  - Furiex Research Site, Loma Linda, California
  - Furiex Research Site, Lomita, California
  - Furiex Research Site, Long Beach, California
  - Furiex Research Site, Los Angeles, California
  - Furiex Research Site, Newport Beach, California
  - Furiex Research Site, North Hollywood, California
  - Furiex Research Site, Northridge, California
  - Furiex Research Site, Pasadena, California
  - Furiex Research Site, Sacramento, California
  - Furiex Research Site, San Diego, California
  - Furiex Research Site, Santa Ana, California
  - Furiex Research Site, Ventura, California
  - Furiex Research Site, Walnut Creek, California
  - Furiex Research Site, Denver, Colorado
  - Furiex Research Site, Boca Raton, Florida
  - Furiex Research Site, Boynton Beach, Florida
  - Furiex Research Site, Bradenton, Florida
  - Furiex Research Site, Brooksville, Florida
  - Furiex Research Site, Clearwater, Florida
  - Furiex Research Site, Cooper City, Florida
  - Furiex Research Site, Coral Springs, Florida
  - Furiex Research Site, Eustis, Florida
  - Furiex Research Site, Fort Lauderdale, Florida
  - Furiex Research Site, Hallandale, Florida
  - Furiex Research Site, Hialeah, Florida
  - Furiex Research Site, Jacksonville, Florida
  - Furiex Research Site, Jupiter, Florida
  - Furiex Research Site, Lauderdale Lakes, Florida
  - Furiex Research Site, Melbourne, Florida
  - Furiex Research Site, Miami, Florida
  - Furiex Research Site, Miramar, Florida
  - Furiex Research Site, New Port Richey, Florida
  - Furiex Research Site, Orlando, Florida
  - Furiex Research Site, Plant City, Florida
  - Furiex Research Site, Port Orange, Florida
  - Furiex Research Site, South Miami, Florida
  - Furiex Research Site, St. Petersburg, Florida
  - Furiex Research Site, Tampa, Florida
  - Furiex Research Site, Wellington, Florida
  - Furiex Research Site, Winter Haven, Florida
  - Furiex Research Site, Winter Park, Florida
  - Furiex Research Site, Alpharetta, Georgia
  - Furiex Research Site, Athens, Georgia
  - Furiex Research Site, Atlanta, Georgia
  - Furiex Research Site, Dunwoody, Georgia
  - Furiex Research Site, Lawrenceville, Georgia
  - Furiex Research Site, Macon, Georgia
  - Furiex Research Site, Marietta, Georgia
  - Furiex Research Site, Norcross, Georgia
  - Furiex Research Site, Savannah, Georgia
  - Furiex Research Site, Stockbridge, Georgia
  - Furiex Research Site, Boise, Idaho
  - Furiex Research Site, Eagle, Idaho
  - Furiex Research Site, Idaho Falls, Idaho
  - Furiex Research Site, Addison, Illinois
  - Furiex Research Site, Chicago, Illinois
  - Furiex Research Site, Evergreen Park, Illinois
  - Furiex Research Site, Hammond, Illinois
  - Furiex Research Site, Springfield, Illinois
  - Furiex Research Site, Brownsburg, Indiana
  - Furiex Research Site, Evansville, Indiana
  - Furiex Research Site, Granger, Indiana
  - Furiex Research Site, Clive, Iowa
  - Furiex Research Site, Pratt, Kansas
  - Furiex Research Site, Shawnee Mission, Kansas
  - Furiex Research Site, Topeka, Kansas
  - Furiex Research Site, Lexington, Kentucky
  - Furiex Research Site, Owensboro, Kentucky
  - Furiex Research Site, Paducah, Kentucky
  - Furiex Research Site, Lake Charles, Louisiana
  - Furiex Research Site, Monroe, Louisiana
  - Furiex Research Site, Hagerstown, Maryland
  - Furiex Research Site, Hollywood, Maryland
  - Furiex Research Site, Boston, Massachusetts
  - Furiex Research Site, Brockton, Massachusetts
  - Furiex Research Site, Watertown, Massachusetts
  - Furiex Research Site, Ann Arbor, Michigan
  - Furiex Research Site, Bay City, Michigan
  - Furiex Research Site, Cadillac, Michigan
  - Furiex Research Site, Grand Rapids, Michigan
  - Furiex Research Site, Kalamazoo, Michigan
  - Furiex Research Site, Troy, Michigan
  - Furiex Research Site, Ypsilanti, Michigan
  - Furiex Research Site, Plymouth, Minnesota
  - Furiex Research Site, Biloxi, Mississippi
  - Furiex Research Site, City of Saint Peters, Missouri
  - Furiex Research Site, Hazelwood, Missouri
  - Furiex Research Site, St Louis, Missouri
  - Furiex Research Site, Billings, Montana
  - Furiex Research Site, Bellevue, Nebraska
  - Furiex Research Site, Elkhorn, Nebraska
  - Furiex Research Site, Lincoln, Nebraska
  - Furiex Research Site, Omaha, Nebraska
  - Furiex Research Site, Las Vegas, Nevada
  - Furiex Research Site, Reno, Nevada
  - Furiex Research Site, Lebanon, New Hampshire
  - Furiex Research Site, Blackwood, New Jersey
  - Furiex Research Site, Edison, New Jersey
  - Furiex Research Site, Elizabeth, New Jersey
  - Furiex Research Site, Marlton, New Jersey
  - Furiex Research Site, Albuquerque, New Mexico
  - Furiex Research Site, Flushing, New York
  - Furiex Research Site, Hollis, New York
  - Furiex Research Site, Mineola, New York
  - Furiex Research Site, New York, New York
  - Furiex Research Site, Chapel Hill, North Carolina
  - Furiex Research Site, Dunn, North Carolina
  - Furiex Research Site, Greensboro, North Carolina
  - Furiex Research Site, Huntersville, North Carolina
  - Furiex Research Site, Kinston, North Carolina
  - Furiex Research Site, Wilmington, North Carolina
  - Furiex Research Site, Winston-Salem, North Carolina
  - Furiex Research Site, Akron, Ohio
  - Furiex Research Site, Beavercreek, Ohio
  - Furiex Research Site, Cincinnati, Ohio
  - Furiex Research Site, Cleveland, Ohio
  - Furiex Research Site, Columbus, Ohio
  - Furiex Research Site, Dayton, Ohio
  - Furiex Research Site, Groveport, Ohio
  - Furiex Research Site, Kettering, Ohio
  - Furiex Research Site, Lima, Ohio
  - Furiex Research Site, Tiffin, Ohio
  - Furiex Research Site, Toledo, Ohio
  - Furiex Research Site, Norman, Oklahoma
  - Furiex Research Site, Oklahoma City, Oklahoma
  - Furiex Research Site, Portland, Oregon
  - Furiex Research Site, Salem, Oregon
  - Furiex Research Site, Carnegie, Pennsylvania
  - Furiex Research Site, Philadelphia, Pennsylvania
  - Furiex Research Site, Pittsburgh, Pennsylvania
  - Furiex Research Site, Scottdale, Pennsylvania
  - Furiex Research Site, Uniontown, Pennsylvania
  - Furiex Research Site, Warwick, Rhode Island
  - Furiex Research Site, Anderson, South Carolina
  - Furiex Research Site, Columbia, South Carolina
  - Furiex Research Site, Easley, South Carolina
  - Furiex Research Site, Mt. Pleasant, South Carolina
  - Furiex Research Site, North Myrtle Beach, South Carolina
  - Furiex Research Site, Rapid City, South Dakota
  - Furiex Research Site, Athens, Tennessee
  - Furiex Research Site, Chattanooga, Tennessee
  - Furiex Research Site, Columbia, Tennessee
  - Furiex Research Site, Jackson, Tennessee
  - Furiex Research Site, Knoxville, Tennessee
  - Furiex Research Site, Smyrna, Tennessee
  - Furiex Research Site, Austin, Texas
  - Furiex Research Site, Beaumont, Texas
  - Furiex Research Site, Bedford, Texas
  - Furiex Research Site, Corsicana, Texas
  - Furiex Research Site, Dallas, Texas
  - Furiex Research Site, Fort Worth, Texas
  - Furiex Research Site, Frisco, Texas
  - Furiex Research Site, Houston, Texas
  - Furiex Research Site, Humble, Texas
  - Furiex Research Site, Hurst, Texas
  - Furiex Research Site, San Antonio, Texas
  - Furiex Research Site, Bountiful, Utah
  - Furiex Research Site, Salt Lake City, Utah
  - Furiex Research Site, West Valley City, Utah
  - Furiex Research Site, Burlington, Vermont
  - Furiex Research Site, Alexandria, Virginia
  - Furiex Research Site, Christiansburg, Virginia
  - Furiex Research Site, Midlothian, Virginia
  - Furiex Research Site, Norfolk, Virginia
  - Furiex Research Site, Richmond, Virginia
  - Furiex Research Site, Charleston, West Virginia
  - Furiex Research Site, Monroe, Wisconsin
- Canada (10):
  - Furiex Research Site, Kelowna, British Columbia
  - Furiex Research Site, St. John's, Newfoundland and Labrador
  - Furiex Research Site, Burlington, Ontario
  - Furiex Research Site, Greater Sudbury, Ontario
  - Furiex Research Site, Hawkesbury, Ontario
  - Furiex Research Site, London, Ontario
  - Furiex Research Site, Newmarket, Ontario
  - Furiex Research Site, Sarnia, Ontario
  - Furiex Research Site, Toronto, Ontario
  - Furiex Research Site, Vaughan, Ontario
- Furiex Research Site, San Juan, Puerto Rico
- United Kingdom (10):
  - Furiex Research Site, Chestfield, Kent
  - Furiex Research Site, Blackpool, Lancashire
  - Furiex Research Site, Birmingham
  - Furiex Research Site, County Durham
  - Furiex Research Site, Coventry
  - Furiex Research Site, Durham
  - Furiex Research Site, Edinburgh
  - Furiex Research Site, Manchester
  - Furiex Research Site, Sheffield
  - Furiex Research Site, Wigan

REFERENCES:
- [Derived] Fant RV, Henningfield JE, Cash BD, Dove LS, Covington PS. Eluxadoline Demonstrates a Lack of Abuse Potential in Phase 2 and 3 Studies of Patients With Irritable Bowel Syndrome With Diarrhea. Clin Gastroenterol Hepatol. 2017 Jul;15(7):1021-1029.e6. doi: 10.1016/j.cgh.2017.01.026. Epub 2017 Feb 3. PMID 28167156
- [Derived] Lembo AJ, Lacy BE, Zuckerman MJ, Schey R, Dove LS, Andrae DA, Davenport JM, McIntyre G, Lopez R, Turner L, Covington PS. Eluxadoline for Irritable Bowel Syndrome with Diarrhea. N Engl J Med. 2016 Jan 21;374(3):242-53. doi: 10.1056/NEJMoa1505180. PMID 26789872

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 3356 participants were prescreened and entered into interactive voice response system for participation in the study. 1146 participants were randomized. One participant was unintentionally randomized twice and was assigned 2 different participant identification numbers due to participant trying to participate at more than 1 study center at once.
Groups:
- Eluxadoline 75 mg: Eluxadoline 75 mg tablets, orally, twice daily for up to 26 weeks treatment period followed by placebo orally, twice daily for next 4 weeks of blinded-placebo period.
- Eluxadoline 100 mg: Eluxadoline 100 mg tablets, orally, twice daily for up to 26 weeks treatment period followed by placebo orally, twice daily for next 4 weeks of blinded-placebo period.
- Placebo: Eluxadoline placebo matching tablets, orally, twice daily for up to 26 weeks treatment period followed by placebo orally, twice daily for next 4 weeks of blinded-placebo period.
Period: Overall Study
Arm/Group | Eluxadoline 75 mg | Eluxadoline 100 mg | Placebo
Started | 381 | 383 | 382
Attended Week 12 Visit | 296 | 301 | 312
Attended Week 26 Visit | 259 | 271 | 278
Participated in Blinded-Placebo Period | 246 | 253 | 272
Completed | 250 | 264 | 273
Not Completed | 131 | 119 | 109
Not completed — Protocol Violation | 0 | 2 | 0
Not completed — Voluntarily withdrew | 70 | 66 | 74
Not completed — Adverse event or SAE | 32 | 28 | 19
Not completed — Physician decision: other | 10 | 8 | 7
Not completed — Lost to Follow-up | 11 | 5 | 6
Not completed — Sponsor decision, specify | 7 | 5 | 0
Not completed — Physician decision: lack of efficacy | 1 | 5 | 3

BASELINE CHARACTERISTICS:
Population: Enrolled set included all participants who were randomized.
Groups:
- Total: Total of all reporting groups
Arm/Group | Eluxadoline 75 mg | Eluxadoline 100 mg | Placebo | Total
Number analyzed (Participants) | 381 | 383 | 382 | 1146
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.0 (13.17) | 45.7 (13.31) | 47.1 (13.82) | 45.9 (13.45)
Age, Customized [Count of Participants; unit: Participants]
  18-40 years | 139 | 146 | 133 | 418
  41-64 years | 206 | 198 | 198 | 602
  ≥65 years | 36 | 39 | 51 | 126
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 261 | 257 | 250 | 768
  Male | 120 | 126 | 132 | 378

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Were Composite Responders Based on Improvements From Baseline in Daily Worst Abdominal Pain and Daily Stool Consistency Scores
Description: Composite responders were defined as participants who met the daily response criteria for at least 50% of the days with diary entries during the interval of interest. A participant must had met both of the following criteria on a given day to be a daily responder: 1) Daily pain response: worst abdominal pain scores in the past 24 hours improved by ≥30% compared to baseline (average of daily worst abdominal pain the week prior to randomization). 2) Daily stool consistency response: Bristol Stool Scale (BSS) score <5 (ie, score of 1, 2, 3, or 4) or the absence of a bowel movement if accompanied by ≥30% improvement in worst abdominal pain compared to baseline pain. Bristol stool scale was defined as 7-point Scale in which a score of 1 = separate hard lumps, 2 = sausage shaped but lumpy, 3 = sausage-like with cracks on the surface, 4 = sausage-like but smooth and soft, 5 = soft blobs with clear cut edges, 6 = fluffy pieces with ragged edges, and 7 = watery with no solid pieces.
Time Frame: Up to 12 weeks
Population: Intention-to-treat (ITT) analysis set included all participants who were randomized into a treatment group and presents data for participants according to their randomization assignment.
Measure: Number; unit: percentage of participants
Arm/Group | Eluxadoline 75 mg | Eluxadoline 100 mg | Placebo
Number analyzed (Participants) | 381 | 382 | 382
percentage of participants | 28.9 | 29.6 | 16.2
Statistical Analysis 1: Comparison: Eluxadoline 75 mg vs Placebo; The family-wise error rate was controlled by Bonferroni adjustment for each active dose versus placebo; Test type: Superiority; p < 0.001, Chi-square test statistic — Significance level of 0.025
Statistical Analysis 2: Comparison: Eluxadoline 100 mg vs Placebo; The family-wise error rate was controlled by Bonferroni adjustment for each active dose versus placebo; Test type: Superiority; p < 0.001, Chi-square test statistic — Significance level of 0.025

2. Secondary Outcome: Percentage of Participants Who Were Composite Responders Based on Improvements From Baseline in Daily Worst Abdominal Pain and Daily Stool Consistency Scores
Description: as for outcome 1
Time Frame: Up to 26 weeks
Population: ITT analysis set included all participants who were randomized into a treatment group and presents data for participants according to their randomization assignment.
Measure: Number; unit: percentage of participants
Arm/Group | Eluxadoline 75 mg | Eluxadoline 100 mg | Placebo
Number analyzed (Participants) | 381 | 382 | 382
percentage of participants | 30.4 | 32.7 | 20.2
Statistical Analysis 1: Comparison: Eluxadoline 75 mg vs Placebo; The family-wise error rate was controlled by Bonferroni adjustment for each active dose versus placebo; Test type: Superiority; p = 0.001, Chi-square test statistic — Significance level of 0.025
Statistical Analysis 2: Comparison: Eluxadoline 100 mg vs Placebo; The family-wise error rate was controlled by Bonferroni adjustment for each active dose versus placebo; Test type: Superiority; p < 0.001, Chi-square test statistic — Significance level of 0.025

3. Secondary Outcome: Percentage of Participants Who Were Pain Responders In Daily Worst Abdominal Pain Scores by Intervals
Description: Pain responders were defined as participants who met the daily pain response criteria (ie, the worst abdominal pain score in the past 24 hours improved by ≥30% compared to baseline) for at least 50% of days with diary entries during each interval. A participant must have had a minimum of 20 days of diary entries over any 4-week interval, a minimum of 60 days of diary entries over the 12-week interval, and a minimum of 110 days of diary entries over the 26-week interval to be a responder.
Time Frame: 12-week interval (Weeks 1-12), 26-week interval (Weeks 1-26), and 4-week interval (Weeks 1-4, 5-8, 9-12, 13-16, 17-20, and 21-24)
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Eluxadoline 75 mg | Eluxadoline 100 mg | Placebo
Number analyzed (Participants) | 381 | 382 | 382
percentage of participants
  Responders during Weeks 1-12 | 48.0 | 51.0 | 45.3
  Responders during Weeks 1-26 | 47.5 | 50.0 | 44.8
  Responders during Weeks 1-4 | 46.7 | 46.6 | 41.9
  Responders during Weeks 5-8 | 53.0 | 52.9 | 49.2
  Responders during Weeks 9-12 | 48.0 | 50.3 | 46.9
  Responders during Weeks 13-16 | 47.2 | 49.0 | 43.5
  Responders during Weeks 17-20 | 45.1 | 47.4 | 42.7
  Responders during Weeks 21-24 | 41.7 | 46.9 | 40.6

4. Secondary Outcome: Percentage of Participants Who Were Responders In Daily Stool Consistency Scores by Intervals
Description: Stool consistency responders: Participants who met daily stool consistency response criterion (ie,score of 1, 2, 3, or 4 or absence of bowel movement if accompanied by ≥30% improvement in worst abdominal pain compared to baseline pain) for at least 50% of days with diary entries during each interval. BSS was defined as 7-point Scale in which score of 1= separate hard lumps, 2= sausage shaped but lumpy, 3= sausage-like with cracks on the surface, 4= sausage-like but smooth and soft, 5= soft blobs with clear cut edges, 6= fluffy pieces with ragged edges, and 7= watery with no solid pieces. A participant must have had a minimum of 20 days of diary entries over any 4-week interval, a minimum of 60 days of diary entries over 12-week interval, and a minimum of 110 days of diary entries over 26-week interval to be a responder.
Time Frame: as for outcome 3
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Eluxadoline 75 mg | Eluxadoline 100 mg | Placebo
Number analyzed (Participants) | 381 | 382 | 382
percentage of participants
  Responders during Weeks 1-12 | 37.0 | 35.6 | 20.9
  Responders during Weeks 1-26 | 34.4 | 39.8 | 23.6
  Responders during Weeks 1-4 | 34.6 | 37.2 | 18.1
  Responders during Weeks 5-8 | 37.5 | 38.2 | 23.3
  Responders during Weeks 9-12 | 37.5 | 39.3 | 26.4
  Responders during Weeks 13-16 | 36.2 | 41.4 | 24.9
  Responders during Weeks 17-20 | 33.9 | 36.1 | 24.9
  Responders during Weeks 21-24 | 32.5 | 38.2 | 22.8

5. Secondary Outcome: Percentage of Participants Who Were Responders In Irritable Bowel Syndrome, Diarrhea Predominant (IBS-d) Global Symptom Scale by Intervals
Description: IBS-d global symptom responders were defined as those participants who met the daily IBS-d global symptom response criteria (ie, IBS-d global symptom score of 0 [none] or 1 [mild]; or a daily IBS-d global symptom score improved by ≥2.0 compared to the baseline average) for at least 50% of days with diary entries during each interval. IBS-d Global Symptom Scale was a 5-point scale, score ranging from 0 to 4. 0= no symptoms, 1= mild symptoms, 2= moderate symptoms, 3= severe symptoms and 4 = very severe symptoms. A participant must have had a minimum of 20 days of diary entries over any 4-week interval, a minimum of 60 days of diary entries over the 12-week interval, and a minimum of 110 days of diary entries over the 26-week interval to be a responder.
Time Frame: as for outcome 3
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Eluxadoline 75 mg | Eluxadoline 100 mg | Placebo
Number analyzed (Participants) | 381 | 382 | 382
percentage of participants
  Responders during Weeks 1-12 | 43.6 | 42.4 | 29.6
  Responders during Weeks 1-26 | 45.1 | 43.2 | 34.3
  Responders during Weeks 1-4 | 40.2 | 36.9 | 25.7
  Responders during Weeks 5-8 | 45.1 | 45.0 | 35.1
  Responders during Weeks 9-12 | 44.9 | 43.5 | 34.0
  Responders during Weeks 13-16 | 43.8 | 42.9 | 33.0
  Responders during Weeks 17-20 | 42.5 | 40.8 | 33.2
  Responders during Weeks 21-24 | 41.7 | 41.6 | 33.8

6. Secondary Outcome: Percentage of Participants Who Were Responders to the Irritable Bowel Syndrome Quality of Life Measure (IBS-QoL) Scale
Description: IBS-QoL responders were defined as participants who achieved at least a 14-point improvement in IBS-QoL total score from baseline to the applicable visit. The IBS-QoL consists of 34 items each with a 5-point response scale, where 1 generally represents better responses on items and 5 represents worse responses. The individual responses to the answered items were summed and standardized for a total score and then transformed to a 0- to 100-point (0= worst; 100=better) scale for ease of interpretation.
Time Frame: Weeks 4, 8, 12, 18, 26 and 30 (End of Treatment [EOT])
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Eluxadoline 75 mg | Eluxadoline 100 mg | Placebo
Number analyzed (Participants) | 381 | 382 | 382
percentage of participants
  Responders at Week 4 | 45.1 | 45.5 | 40.1
  Responders at Week 8 | 48.8 | 50.0 | 43.7
  Responders at Week 12 | 48.3 | 49.5 | 45.0
  Responders at Week 18 | 45.1 | 45.0 | 41.9
  Responders at Week 26 | 45.4 | 44.8 | 41.4
  Responders at Week 30 /EOT | 54.3 | 53.9 | 52.6

7. Secondary Outcome: Percentage of Participants With Irritable Bowel Syndrome - Adequate Relief (IBS-AR) Scale
Description: Adequate relief of IBS symptoms was assessed once weekly by participants answering the IBS-AR item in the electronic diary. IBS-AR responders were defined as participants with a weekly response of "Yes" to adequate relief of their IBS symptoms for at least 50% of the total weeks during the interval. A participant must have had a positive response on ≥6 weeks for the 12-week interval and ≥13 weeks for the 26-week interval, regardless of diary compliance, to be a responder.
Time Frame: 12-week interval (Weeks 1-12) and 26-week interval (Weeks 1-26)
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Eluxadoline 75 mg | Eluxadoline 100 mg | Placebo
Number analyzed (Participants) | 381 | 382 | 382
percentage of participants
  Responders during Weeks 1-12 | 60.1 | 58.4 | 49.2
  Responders during Weeks 1-26 | 52.8 | 53.7 | 43.7

8. Secondary Outcome: Change From Baseline in Daily Abdominal Discomfort Scores
Description: Symptoms of abdominal discomfort were recorded on a 0 to 10 scale, where 0 corresponded to no discomfort and 10 corresponded to worst imaginable discomfort. A negative change from Baseline indicates the discomfort decreased.
Time Frame: Baseline, Weeks 4, 12 and 26
Population: ITT analysis set included all participants who were randomized into a treatment group and presents data for participants according to their randomization assignment. Here, number analyzed is the participants who were evaluable at specific time point.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Eluxadoline 75 mg | Eluxadoline 100 mg | Placebo
Number analyzed (Participants) | 381 | 382 | 382
score on a scale
  Change at Week 4: number analyzed (Participants) | 348 | 351 | 364
  Change at Week 4 | -2.44 (2.219) | -2.19 (2.120) | -2.06 (2.063)
  Change at Week 12: number analyzed (Participants) | 298 | 303 | 316
  Change at Week 12 | -2.88 (2.417) | -2.90 (2.175) | -2.56 (2.461)
  Change at Week 26: number analyzed (Participants) | 255 | 267 | 267
  Change at Week 26 | -3.19 (2.454) | -3.16 (2.362) | -2.76 (2.582)

9. Secondary Outcome: Change From Baseline in Daily Abdominal Bloating Scores
Description: Symptoms of abdominal bloating were recorded on a 0 to 10 scale, where 0 corresponded to no bloating and 10 corresponded to worst imaginable bloating. A negative change from Baseline indicates the bloating decreased.
Time Frame: Baseline, Weeks 4, 12 and 26
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Eluxadoline 75 mg | Eluxadoline 100 mg | Placebo
Number analyzed (Participants) | 381 | 382 | 382
score on a scale
  Change at Week 4: number analyzed (Participants) | 292 | 305 | 302
  Change at Week 4 | -1.89 (2.170) | -1.80 (2.204) | -1.73 (2.081)
  Change at Week 12: number analyzed (Participants) | 247 | 262 | 259
  Change at Week 12 | -2.24 (2.445) | -2.41 (2.396) | -2.08 (2.492)
  Change at Week 26: number analyzed (Participants) | 210 | 229 | 214
  Change at Week 26 | -2.38 (2.619) | -2.68 (2.673) | -2.17 (2.682)

10. Secondary Outcome: Number of Bowel Movements Per Day
Description: Participants recorded the number of bowel movements over 24 hours daily throughout the treatment.
Time Frame: Weeks 4, 12 and 26
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: bowel movements per day
Arm/Group | Eluxadoline 75 mg | Eluxadoline 100 mg | Placebo
Number analyzed (Participants) | 381 | 382 | 382
bowel movements per day
  Week 4: number analyzed (Participants) | 348 | 351 | 364
  Week 4 | 3.03 (2.021) | 3.05 (1.962) | 3.38 (1.856)
  Week 12: number analyzed (Participants) | 298 | 303 | 316
  Week 12 | 2.89 (2.057) | 2.80 (1.685) | 3.15 (1.991)
  Week 26: number analyzed (Participants) | 255 | 267 | 267
  Week 26 | 2.57 (1.637) | 2.66 (1.625) | 2.96 (1.931)

11. Secondary Outcome: Number of Bowel Incontinence Episodes
Description: Participants recorded the number of incontinence episodes over 24 hours daily throughout the treatment.
Time Frame: Weeks 4, 12 and 26
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: incontinence episodes
Arm/Group | Eluxadoline 75 mg | Eluxadoline 100 mg | Placebo
Number analyzed (Participants) | 381 | 382 | 382
incontinence episodes
  Week 4: number analyzed (Participants) | 348 | 351 | 364
  Week 4 | 0.47 (1.304) | 0.41 (1.230) | 0.50 (1.195)
  Week 12: number analyzed (Participants) | 298 | 303 | 316
  Week 12 | 0.40 (1.083) | 0.28 (0.875) | 0.46 (1.269)
  Week 26: number analyzed (Participants) | 255 | 267 | 267
  Week 26 | 0.30 (0.982) | 0.27 (0.844) | 0.50 (1.503)

12. Secondary Outcome: Number of Bowel Incontinence Free Days
Description: An incontinence free day was one where the participant reports zero incontinence episodes. The number of incontinence free days for a participant was assessed each week based on the number of reported days.
Time Frame: Weeks 4, 12 and 26
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Eluxadoline 75 mg | Eluxadoline 100 mg | Placebo
Number analyzed (Participants) | 381 | 382 | 382
days
  Week 4: number analyzed (Participants) | 348 | 351 | 364
  Week 4 | 5.53 (2.282) | 5.46 (2.264) | 5.31 (2.444)
  Week 12: number analyzed (Participants) | 298 | 303 | 316
  Week 12 | 5.38 (2.320) | 5.56 (2.164) | 5.28 (2.364)
  Week 26: number analyzed (Participants) | 255 | 267 | 267
  Week 26 | 5.53 (2.129) | 5.59 (2.216) | 5.29 (2.322)

13. Secondary Outcome: Number of Urgency Episodes Per Day
Description: Participants recorded the number of urgency episodes over 24 hours daily throughout the treatment.
Time Frame: Weeks 4, 12 and 26
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: episodes per day
Arm/Group | Eluxadoline 75 mg | Eluxadoline 100 mg | Placebo
Number analyzed (Participants) | 381 | 382 | 382
episodes per day
  Week 4: number analyzed (Participants) | 348 | 351 | 364
  Week 4 | 1.62 (1.948) | 1.58 (1.732) | 2.00 (1.779)
  Week 12: number analyzed (Participants) | 298 | 303 | 316
  Week 12 | 1.37 (1.884) | 1.32 (1.675) | 1.73 (1.785)
  Week 26: number analyzed (Participants) | 255 | 267 | 267
  Week 26 | 1.13 (1.580) | 1.12 (1.576) | 1.54 (1.826)

14. Secondary Outcome: Change From Baseline in IBS-QoL Total Scores
Description: The IBS-QoL consists of 34 items each with a 5-point response scale, where 1 generally represents better responses on items and 5 represents worse responses. The individual responses to the answered items were summed and standardized for a total score and then transformed to a 0- to 100- point scale (0=worst; 100=better) for ease of interpretation. A positive change from Baseline indicates that quality of life improved.
Time Frame: Baseline, Weeks 4, 8, 12, 18, 26 and 30/EOT
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Eluxadoline 75 mg | Eluxadoline 100 mg | Placebo
Number analyzed (Participants) | 381 | 382 | 382
score on a scale
  Change at Week 4: number analyzed (Participants) | 335 | 342 | 357
  Change at Week 4 | 17.51 (19.755) | 17.26 (18.980) | 14.07 (18.787)
  Change at Week 8: number analyzed (Participants) | 318 | 319 | 333
  Change at Week 8 | 21.60 (20.762) | 21.10 (21.925) | 16.62 (20.856)
  Change at Week 12: number analyzed (Participants) | 293 | 300 | 311
  Change at Week 12 | 22.69 (21.723) | 22.62 (24.017) | 19.50 (21.636)
  Change at Week 18: number analyzed (Participants) | 275 | 281 | 293
  Change at Week 18 | 24.17 (22.761) | 23.52 (24.029) | 20.64 (23.268)
  Change at Week 26: number analyzed (Participants) | 258 | 271 | 277
  Change at Week 26 | 24.91 (22.638) | 24.19 (24.599) | 21.50 (23.709)
  Change at Week 30/EOT: number analyzed (Participants) | 335 | 344 | 342
  Change at Week 30/EOT | 22.79 (22.329) | 20.92 (23.724) | 21.63 (23.376)

ADVERSE EVENTS:
Time Frame: From first dose of study drug up to 30 weeks
Description: Safety Set: all participants who received at least 1 dose of drug per actual treatment received. 1 participant in 100 mg arm received 75 mg, 2 participants in Placebo arm received eluxadoline 75 mg and 100 mg. AEs for each period were analyzed separately. In the Other AE section, a result of 0 in an arm means the ≥5% threshold was not met.
Groups:
- Eluxadoline 75 mg (Treatment Period): Eluxadoline 75 mg tablets, orally, twice daily for up to 26 weeks period.
- Eluxadoline 100 mg (Treatment Period): Eluxadoline 100 mg tablets, orally, twice daily for up to 26 weeks period.
- Placebo (Treatment Period): Eluxadoline placebo matching tablets, orally, twice daily for up to 26 weeks period.
- Eluxadoline 75 mg (Blinded-Placebo Period): Participants who received eluxadoline 75 mg in treatment period were administered with placebo orally, twice daily for next 4 weeks.
- Eluxadoline 100 mg (Blinded-Placebo Period): Participants who received eluxadoline 100 mg in treatment period were administered with placebo orally, twice daily for next 4 weeks.
- Placebo (Blinded-Placebo Period): Participants who received placebo matching tablets in treatment period were administered with placebo orally, twice daily for next 4 weeks.
Arm/Group | Eluxadoline 75 mg (Treatment Period) | Eluxadoline 100 mg (Treatment Period) | Placebo (Treatment Period) | Eluxadoline 75 mg (Blinded-Placebo Period) | Eluxadoline 100 mg (Blinded-Placebo Period) | Placebo (Blinded-Placebo Period)
All-Cause Mortality (participants affected / at risk) | 0/379 | 0/380 | 0/381 | 0/246 | 0/253 | 0/272
Serious Adverse Events (participants affected / at risk) | 9/379 | 14/380 | 8/381 | 0/246 | 0/253 | 0/272
Other Adverse Events (participants affected / at risk) | 97/379 | 97/380 | 69/381 | 0/246 | 0/253 | 0/272
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Eluxadoline 75 mg (Treatment Period) (N=379) | Eluxadoline 100 mg (Treatment Period) (N=380) | Placebo (Treatment Period) (N=381) | Eluxadoline 75 mg (Blinded-Placebo Period) (N=246) | Eluxadoline 100 mg (Blinded-Placebo Period) (N=253) | Placebo (Blinded-Placebo Period) (N=272)
Abdominal discomfort (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Colitis ischemic (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Gastric ulcer (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Hiatus hernia (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Pancreatitis acute (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 0 | 0
Umbilical hernia (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Appendicitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Bacterial pyelonephritis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Enterocolitis infections (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Liver abscess (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Pyelonephritis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Chest pain (General disorders) | 1 | 1 | 0 | 0 | 0 | 0
Non-cardiac pain (General disorders) | 0 | 1 | 0 | 0 | 0 | 0
Acute coronary syndrome (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0
Angina pectoris (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0
Coronary artery disease (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0
Headache (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Myasthenia gravis (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Hepatitis (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0 | 0
Concussion (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0
Pseudomeningocele (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0
ECG T wave abnormal (Investigations) | 0 | 1 | 0 | 0 | 0 | 0
Hepatic enzyme increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Suicide attempt (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0
Dysfunctional uterine bleeding (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0 | 0
Ovarian cyst ruptured (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0 | 0
Uterine prolapse (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Eluxadoline 75 mg (Treatment Period) (N=379) | Eluxadoline 100 mg (Treatment Period) (N=380) | Placebo (Treatment Period) (N=381) | Eluxadoline 75 mg (Blinded-Placebo Period) (N=246) | Eluxadoline 100 mg (Blinded-Placebo Period) (N=253) | Placebo (Blinded-Placebo Period) (N=272)
Constipation (Gastrointestinal disorders) | 33 | 30 | 8 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 31 | 33 | 22 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 19 | 13 | 15 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 13 | 22 | 17 | 0 | 0 | 0
Headache (Nervous system disorders) | 14 | 23 | 22 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor will work with the Investigators to determine how any manuscript or publication in a scientific journal is written and edited, the number and order of authors, the publication to which it will be submitted, and other related issues. The sponsor has final approval authority over all such issues. Data are the property of the sponsor and cannot be published without prior authorization from the sponsor, but data and publication thereof will not be unduly withheld.